CLINICAL TRIAL: NCT06412510
Title: Prehabilitation for Elderly Patients With Advanced Epithelial Ovarian, Fallopian Tube, Primary Peritoneal Carcinoma and Pancreatic Cancer Undergoing Neoadjuvant Chemotherapy
Brief Title: Prehabilitation for EOC, Fallopian Tube, Primary Peritoneal Carcinoma and Pancreatic Cancer w/ NACT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE3824
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Cancer; Epithelial Ovarian Cancer; Pancreatic Adenocarcinoma
Keywords: Ovarian Cancer; Neoadjuvant chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Arm 1 (Experimental): Exercise Intervention: Participants will be referred to Langston Hughes Community Center and work with exercise physiologists who will utilize our SmartGym ecosystem in providing exercise assessments, prescriptions, and training.
  Nitrition Intervention: Participants in the intervention group will be provided with 1-2 bottles of high protein oral nutritional supplements daily (ONS) to ensure that protein needs are met daily. There will be two options of ONS to choose from: one option a high calorie, high protein supplement, and the other option a low fat/low sugar, high protein supplement.
  Supportive care/Mind-body intervention: Participants will have access to Taussig Cancer Institute Patient Support services that are offered for free.
  Interventions: Other: Prehabilitation
- Control - Arm 2 (No Intervention): Exercise: Standard of care. Level of activity will be reported and monitored at each visit through study coordinator assessment and patient interview.
  Nutrition: Participants will be referred to dietitian and will be seen for a baseline evaluation, as needed throughout treatment and post treatment. A full nutrition assessment will be performed, and malnutrition diagnosis will be documented. When no malnutrition is identified participants will be provided general nutrition counseling related to their cancer type, cancer treatment, and recommendations for symptom management as needed. Those participants identified to be malnourished to any degree will receive personalized medical nutrition therapy including nutrition interventions to improve caloric intake.
  Supportive care/Mind-body intervention: Per standard of care, participants will be offered support services from Taussig Cancer Institute program.

INTERVENTIONS:
Other: Prehabilitation — Exercise Intervention: SmartGyms, band or smartphone used to scan into the TechnoGym MyWellness kiosk, which controls the TechnoGym Excite Live and Biostrength equipment. The exercise session will consist of a program that adheres to the FITT (Frequency, Intensity, Timing, and Type) exercise prescription in accordance with ACSM 2018 ACSM Roundtable recommendations for Physical Function for combined Aerobic and Resistance training.
  Nutrition Intervention: 30 gm protein supplement
  Supportive care/Mind-body intervention: Yoga, mindfulness practices, art therapy, and music therapy
  Arms: Intervention - Arm 1

SUMMARY:
The purpose of this study is to see whether participants who are assigned to a multimodal prehabilitation intervention during chemotherapy are able to adhere with exercise and nutrition program to prepare for their cancer surgery.

DETAILED DESCRIPTION:
Elderly participants with epithelial ovarian cancer (EOC) and pancreatic adenocarcinoma (PDAC) undergoing neoadjuvant chemotherapy (NACT) are often frail and malnourished. Both chemotherapy and disease burden are associated with a decline in muscle mass leading to decrease in physical strength and cardiovascular fitness. Limited efforts have focused on decreasing morbidity at time of chemotherapy and surgery and improving functional capacity. Exercise during chemotherapy has been shown to improve chemotherapy related symptoms and quality of life in participants with breast cancer participants. In surgical patient populations, preoperative rehabilitation (prehabilitation) has been shown to improve walking capacity, decrease hospital length of stay, perioperative complications, and cost. However, whether multimodal prehabilitation improves the functional capacity and perioperative outcomes of EOC and PDAC participants undergoing NACT compared to standard of care is unknown. Investigators aim to evaluate if prehabilitation in participants with EOC and PDAC undergoing NACT improves physical fitness/ functional outcomes, perioperative outcomes, nutritional status, and quality of life compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and older
* Patients with diagnosis of advanced (Stage III or IV) epithelial ovarian, fallopian tube, or
* Patients with diagnosis of pancreatic adenocarcinoma (PDAC) (Stage I, II, or III) undergoing neoadjuvant chemotherapy.
* Patients with locally advanced esophageal cancer undergoing neoadjuvant chemotherapy.
* Patients with locally advanced muscle invasive bladder cancer undergoing neoadjuvant chemotherapy.

Exclusion Criteria:

* Life expectancy less than 3 months in the opinion of the treating physician
* Patients unable to provide informed consent.
* Wheelchair bound patients/ physical immobility.
* Severe cardiopulmonary disease defined as NYHA class III or IV
* Patients with malignant bowel obstruction who will require surgical intervention or nutritional support in the form of enteral or parenteral nutrition will also be excluded.
* Patients with any other comorbidity or condition, which, in the opinion of the enrolling investigator, would place the patient at unnecessarily higher greater risk or burden, or participating in the study would not be in the best interests of the patient.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Rate of adherence as calculated by the compliance percentage | 6 weeks post intervention
  Compliance will be defined as completion of at least 2 exercise sessions per week (75%) for the duration of the study.

SECONDARY OUTCOMES:
Change in effectiveness of prehabilitation as assessed by 1 Rep Max Isokinetic strength test | Baseline, 6 weeks post intervention
  Rep Max Isokinetic Strength Test measured by BiostrengthTM Maximal Strength
Change in effectiveness of prehabilitation as assessed by Grade Exercise Test Grade Exercise Test measured by Grade Exercise Test. | Baseline, 6 weeks post intervention
  At baseline, and within the immediate post-exercise recovery, rating of perceived exertion (RPE; Borg scale, 6-20) will be assessed. Peak exercise exhaustion was verified if two or more of the following criteria were met: 1)96 HR within 10 bpm of age-predicted maximum HR (220-age), 2) RPE > 17, and/or 3) a plateau in HR (<3 bpm change over the last two intensity stages).
  VO2 max will be calculated by ACSM's Treadmill Walking Equation:
  VO2 [ml/kg/min] = (0.1 x speed) + (1.8 x Speed x Grade) 3.5 ml/kg/min
Change in effectiveness of prehabilitation as assessed by timed up and go test | Baseline, 6 weeks post intervention
  Timed up and go test is one unit of time to measure how fast patients can move
Change in effectiveness of prehabilitation as assessed by grip strength test | Baseline, 6 weeks post intervention
  Grip strength test measured by handheld dynamometer
Change in effectiveness of prehabilitation as assessed by 30 second sit to stand test | Baseline, 6 weeks post intervention
  The number of times a patient can rise to a standing position from a seated position without the use of their upper extremities is counted in a thirty second period.
Change in measure of balance as assessed by unipedal stance test | Baseline, 6 weeks post intervention
  This is a measure of balance and is assessed by asking the participant to stand on one foot (of their choice) with the lifted foot remaining close to their opposite ankle, first with eyes open and then with eyes closed.The amount of time a participant can stand on one foot is recorded.
Effectiveness of prehabilitation as assessed by measuring the change in body mass composition | Baseline, 6 weeks post-intervention
  Body composition measured using contrast-enhanced CT scan
Effectiveness of prehabilitation as assessed by the change in nutritional status | Baseline, Cycle 2 day 1, cycle 3 day 1, cycle 4 day 1(each cycle is 21 days) and 6 weeks post-intervention
  Assessed for the presence of malnutrition per the Cleveland Clinic organization's standard of care based on American Society for Parenteral and Enteral Nutrition (ASPEN) and the Academy of Nutrition and Dietetics (AND) (ASPEN/AND) guidelines, and by assessing changes in the degree of malnutrition throughout the study period
Quality of life as assessed by FACT-G7 (Functional Assessment of Cancer Therapy) | At baseline
  Functional Assessment of Cancer Therapy(FACT-G7) to assess the illness is measured on a scale from 0 to 4, where 0 is 'not at all' and 4 is 'very much'
Quality of life as assessed by FACT-G7 (Functional Assessment of Cancer Therapy) | Up to 6 weeks post intervention
  Functional Assessment of Cancer Therapy(FACT-G7) to assess the illness is measured on a scale from 0 to 4, where 0 is 'not at all' and 4 is 'very much'
Quality of life as assessed by FACT-O | At baseline
  FACT-O to assess the illness is measured on a scale from 0 to 4, where 0 is 'not at all' and 4 is 'very much'
Quality of life as assessed by FACT-O | Up to 6 weeks post intervention
  FACT-O to assess the illness is measured on a scale from 0 to 4, where 0 is 'not at all' and 4 is 'very much'
Effectiveness of prehabilitation as assessed by Chemotherapy toxicity | At cycle 2, day 1(each cycle is 21 days)
  Chemotherapy toxicity as measured by the standard CTCAE v5 grading system
Effectiveness of prehabilitation as assessed by Chemotherapy toxicity | At cycle 3, day 1(each cycle is 21 days)
  Chemotherapy toxicity as measured by the standard CTCAE v5 grading system
Effectiveness of prehabilitation as assessed by Chemotherapy toxicity | At cycle 4, day 1(each cycle is 21 days)
  Chemotherapy toxicity as measured by the standard CTCAE v5 grading system
Effectiveness of prehabilitation as assessed by Chemotherapy toxicity | Up to 6 weeks post intervention
  Chemotherapy toxicity as measured by the standard CTCAE v5 grading system
Effectiveness of prehabilitation as assessed by participant acceptability of intervention survey using IAM(Intervention appropriateness measure) | Up to 6 weeks post intervention
  IAM is measured on a scale of 1 to 5, where 1 is completely disagree and 5 is completely agree.
Effectiveness of prehabilitation as assessed by participant acceptability of intervention survey using FIM(Feasibility of intervention measure) | Up to 6 weeks post intervention
  FIM is measured on a scale of 1 to 5, where 1 is completely disagree and 5 is completely agree.
Effectiveness of prehabilitation as assessed by participant acceptability scale | Baseline
  Participant acceptability of anxiety and depression screening as measured by Hospital anxiety and depression scale(HADS) scoring from 0-21 where 0-7 is normal;8-10 is borderline abnormal; 11-21 is abnormal
Effectiveness of prehabilitation as assessed by participant acceptability scale | Up to 6 weeks post intervention
  Participant acceptability of anxiety and depression screening as measured by Hospital anxiety and depression scale(HADS) scoring from 0-21 where 0-7 is normal;8-10 is borderline abnormal; 11-21 is abnormal

CONTACTS AND LOCATIONS:
Overall Officials: Mariam AlHilli, MD, Principal Investigator — Cleveland Clinic Foundation, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication will be shared with scientific journals during peer-review or at scientific/medical conferences/meetings. All IDP will be anonymized.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available during the course of the study and indefinitely thereafter.
Access Criteria: The data will be available as it pertains to journal publication to the scientific/medical community. This study has no intellectual property data that would require a CDA be in place.